CLINICAL TRIAL: NCT04696406
Title: Multicenter, Multinational, Clinical Trial of the Performance of RESPINOR DXT to Identify Patients at Increased Risk of Weaning Failure
Acronym: DE-RISK WF
Status: Completed | Type: Observational
Sponsor: Respinor AS (Industry)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Other Study IDs: DXT-CS-005
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Failure
Keywords: Diaphragm ultrasound; Diaphragm function; Mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weaning failure: Defined as the failure to pass a spontaneous breathing trial or the need for reintubation or death within 48 hours
  Interventions: Device: RESPINOR DXT
- Weaning success: Defined as a successful spontaneous breathing trial and is not reintubated or dies in the first 48 hours after extubation.
  Interventions: Device: RESPINOR DXT

INTERVENTIONS:
Device: RESPINOR DXT — Blinded, continuous diaphragmatic excursion measurements by DXT will be conducted during the patients' first SBT. The recording shall be initiated 15 minutes prior to the first SBT and will end 15 minutes post SBT.

SUMMARY:
The study will be a multicenter, multinational, prospective single arm blinded study to validate DXT's performance to identify patients at increased risk of weaning failure during the spontaneous breathing trial (SBT). Continuous diaphragmatic excursion measurements by DXT will be conducted during the patients' first SBT. The recording shall be initiated 15 minutes prior to the first SBT and will end 15 minutes post SBT.

All patients on mechanical ventilation in the ICU meeting the eligibility criteria shall undergo a daily screen for weaning readiness. If any of the components of the daily screen is not met, the patient will not undergo a SBT that day and continued to be screened daily. Patients passing daily screening criteria shall automatically receive an SBT.

The SBT shall last for 30-120 minutes and be performed on continuous positive airway pressure up to 5 cm H2O and pressure support up to 7 cm H2O. The SBT shall be terminated and mechanical ventilation reinstituted at the original settings if the patient meets any of the SBT failure criteria.

A trial is considered successful and physicians will be asked to approve extubation when the patient can breathe spontaneously for the whole trial.

Patients shall be continued to be screened daily until extubation, 21 days after enrolment, performance of tracheostomy, death, or withdrawal of care. All patients shall be followed until hospital discharge or death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and able to give informed consent (either themselves or next of kin)
2. Have undergone invasive mechanical ventilation > 24 hours
3. Ready to wean according to criteria (from the sixth international consensus conference on intensive care medicine):

   1. Adequate cough
   2. Absence of excessive tracheobronchial secretion
   3. Resolution of disease acute phase for which the patient was intubated
   4. Clinical stability, defined as stable cardiovascular status (i.e. fC < 140 beats·min-1, systolic BP 90-160 mmHg, no or minimal vasopressors) and stable metabolic status
   5. Adequate oxygenation, defined as SaO2 > 90% on < FIO2 0.4 (or PaO2/FIO2 > 150 mmHg) and PEEP < 8 cmH2O
   6. Adequate pulmonary function, i.e. fR < 35 breaths·min-1
   7. Adequate mentation, defined as no sedation or adequate mentation on sedation (or stable neurologic patient), i.e., patient awake, calm and responsive to simple orders (squeeze hand, knock the head, close the eyes), no agitation.

Exclusion Criteria:

1. Not registered with a social security system nor entitled to be
2. Central or spinal neurological injury involving central ventilatory control
3. Presence of a neuromuscular disease involving respiratory muscles
4. Use of muscle-paralyzing agents within 24h before the study, except if given for intubation
5. Known paralysis of a hemidiaphragm or suspicion of paralysis of a hemidiaphragm, defined by the radiographic evidence of elevation of a dome > 2.5 cm compared to the contralateral dome
6. Tracheostomy
7. Body mass index >35 kg/m2
8. Patient with therapeutic limitation, i.e. reduced expectancy to survive
9. Pregnant woman or protected adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under invasive mechanical ventilation in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Difference in the rate of weaning failure between patients with a DE < 1.1 cm compared to those with a DE > 1.1 cm. | Second minute of the first SBT
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.1 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RR) statistic will be used to assess the null hypothesis of equality.

SECONDARY OUTCOMES:
Difference in the rate of weaning failure with reintubation failure 72 hours and 7 days after extubation between patients with a DE <1.1 cm compared to those with a DE >1.1 cm. | Second minute of the first SBT
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.1 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RR) statistic will be used to assess the null hypothesis of equality.
Subgroup analysis on the difference in the rate of weaning failure between patients with a DE <1.1 cm compared to those with a DE >1.1 cm excluding COVID-19 patients. Similar subgroup analysis for COVID-19 patients. | Second minute of the first SBT
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.1 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RR) statistic will be used to assess the null hypothesis of equality.
Correlation between median DE measurements taken during the second minute of the SBT and duration of mechanical ventilation prior to the first SBT, after the SBT and total mechanical ventilation time. | Second minute of the first SBT
  Plots of DE values versus MV duration will be presented, together with the estimated correlation coefficient.
Correlation between median DE measurements taken during the second minute of the SBT and duration of ICU stay prior to the first SBT, after the SBT and total ICU time. | Second minute of the first SBT
  Plots of DE values versus ICU duration will be presented, together with the estimated correlation coefficient.
Confirm thresholds for DE to predict weaning outcome during the SBT for the whole sample. | Second minute of the first SBT
  Thresholds for continuous DE will be defined by ROC curve analysis.

OTHER OUTCOMES:
Efficacy - number of patients with overall acceptable signal quality from predefined quality criteria | First SBT
Safety - skin irritation severity | After first SBT, when removing the sensors
  options 'no irritation', slight redness', 'red and moist tissue', 'granulation tissue', and 'infection leading to debridement'
Time spent on achieving good sensor placement | During sensor attachment before the first SBT
  with options 0-5, 6-10 mins, 11-20 mins, 21-30 mins, > 30 mins
Safety - skin irritation frequency | After first SBT, when removing the sensors
  Frequency of skin irritation presented in percentage for each category of skin irritation severity
Criteria for the Earlier Termination of the Trial - sample size calculation based on weaning failure rate | When a minimum of 154 subjects have been enrolled (180 when accounting for dropouts), through study completion, assessed up to 1 year
  Sample size have been calculated with the basis of 4 main assumptions: proportion of weaning failure, assumed relative risk (RR), level of significance, and power. Of these, the proportion of weaning failure is independent of the outcome. Weaning failure rate was assumed to be 20%, requiring 218 patients to meet the endpoints (250 patients accounting for dropouts). If the observed weaning failure is 25%, the number of patients needed is 154 under the same assumptions. One interim assessment of study progress will be conducted. If the observed total proportion of weaning failure is 25% or above (only using the eCRF data, still blinded to the output from DXT), the Sponsor and Principal Investigator can recommend that the trial be concluded and analyzed according to the statistical analysis plan. The interim assessment will be conducted by calculating a 95% CI for the overall weaning failure. The CI will be calculated using the standard normal approximation for one sample proportions.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Demoule, MD, Principal Investigator — Hôpital Universitaire Pitié Salpêtrière; Michele Umbrello, MD, Principal Investigator — Ospedale San Carlo Borromeo; Øyvind Skraastad, MD, Principal Investigator — Oslo University Hospital
Locations (9):
- France (6):
  - Hopital Saint-Antoine, Paris, Cedex 12
  - Hôpitaux Universitaires de Marseille - AP-HM, Marseille, Chem. Des Bourrely
  - Centre Hospitalier Universitaire de Montpellier, Montpellier, Select One...
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hôpital Universitaire Pitié Salpêtrière, Paris
- Ospedale San Carlo Borromeo, Milan, Italy
- Norway (2):
  - Oslo University Hospital, Oslo
  - St. Olavs University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided